CLINICAL TRIAL: NCT05493293
Title: Prospective, Long-Term, Interventional, Active Extension Study to Evaluate the Safety and Tolerability of NBI-921352 as Adjunctive Therapy in Subjects With Focal Onset Seizures (FOS)
Brief Title: Extension Study to Evaluate the Safety and Tolerability of NBI-921352 When Used With Anti-seizure Medications in Adults With Focal Onset Seizures
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The long-term extension study was terminated because the parent study NBI-921352-FOS2021 (NCT05159908) failed to meet its primary endpoint.
Sponsor: Neurocrine Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NBI-921352-FOS2022; 2021-004265-12 (EudraCT Number)
Record Dates: First submitted 2022-08-05; First posted 2022-08-09 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Focal Onset Seizure; Focal Onset Epilepsy
Keywords: epilepsy; focal seizure; sodium channel; voltage-gated; alpha subunit; Nav1.6 inhibitor; antiseizure medicine; ASM; antiepileptic drug; AED; partial seizure; partial onset epilepsy
MeSH Terms: conditions — Seizures; Epilepsy

STUDY DESIGN:
Masking Description: For participants who enroll directly from Study NBI-921352-FOS2021, the study will include a Blinded Dose Conversion Period (1 week) before proceeding to the Open-Label Treatment Period.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- NBI-921352 Treatment (Experimental): Treatment for up to 107 weeks.
  Interventions: Drug: NBI-921352

INTERVENTIONS:
Drug: NBI-921352 — Tablets for oral administration

SUMMARY:
This Phase 2, prospective, interventional, active extension study was designed to evaluate the long-term safety and tolerability of NBI-921352 as adjunctive therapy in adult participants with focal onset seizures who completed 11 weeks of treatment in randomized, double-blind, placebo-controlled Study NBI-921352-FOS2021. Eligible participants may enroll directly following the completion of the Week 11 study visit of Study NBI-921352-FOS2021 or after a gap following completion of that study.

ELIGIBILITY:
Key Inclusion Criteria:

* Provided informed consent.
* Completed 11 weeks of treatment in Study NBI-921352-FOS2021.
* Stable treatment with at least 1 but not more than 4 antiseizure medicines.

Key Exclusion Criteria:

* Have developed any other disorder for which the treatment takes priority over the treatment of focal onset seizure or is likely to interfere with study treatment or impair treatment compliance.

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2022-11-09 (Actual); Primary Completion 2024-03-11 (Actual); Study Completion 2024-03-11 (Actual)

PRIMARY OUTCOMES:
The occurrence of serious treatment-emergent adverse events (TEAEs) | Through Week 111

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Lead, Study Director — Neurocrine Biosciences
Locations (22):
- Australia (3):
  - Neurocrine Clinical Site, Fitzroy
  - Neurocrine Clinical Site, Heidelberg
  - Neurocrine Clinical Site, Melbourne
- Belgium (3):
  - Neurocrine Clinical Site, Brussels
  - Neurocrine Clinical Site, Ghent
  - Neurocrine Clinical Site, Leuven
- Czechia (4):
  - Neurocrine Clinical Site, Brno
  - Neurocrine Clinical Site, Ostrava
  - Neurocrine Clinical Site, Prague
  - Neurocrine Clinical Site, Rychnov nad Kněžnou
- France (4):
  - Neurocrine Clinical Site, Bron
  - Neurocrine Clinical Site, Lille
  - Neurocrine Clinical Site, Rennes
  - Neurocrine Clinical Site, Toulouse
- Hungary (2):
  - Neurocrine Clinical Site, Budapest
  - Neurocrine Clinical Site, Pécs
- Italy (3):
  - Neurocrine Clinical Site, Bologna
  - Neurocrine Clinical Site, Milan
  - Neurocrine Clinical Site, Pavia
- Spain (3):
  - Neurocrine Clinical Site, Barcelona
  - Neurocrine Clinical Site, Madrid
  - Neurocrine Clinical Site, Valencia

IPD SHARING:
Plan to Share IPD: No